CLINICAL TRIAL: NCT03319238
Title: OBSERVATIONAL STUDY OF THE MANAGEMENT OF PATIENTS WITH CHRONIC PAIN
Acronym: OKAPI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-349
Record Dates: First submitted 2017-09-07; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Neuropathic pain; Ketamine; Concomitant treatment; Adverse effect
MeSH Terms: conditions — Chronic Pain; Neuralgia | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient cohort: Neuropathic pain patient taking ketamine
  Interventions: Other: ketamine

INTERVENTIONS:
Other: ketamine — The aim of this study is to evaluate the safety of use, benefits and risks of repeated use of ketamine for each patient with chronic pain in different structures of pain management.

SUMMARY:
The aim of this study is to evaluate the safety of use, benefits and risks of repeated use of ketamine for each patient with chronic pain in different structures of pain management.

DETAILED DESCRIPTION:
This is an observational, longitudinal and multicenter study about use of ketamine. Benefits are assessed with pain intensity, anxiety, depression, quality of life and global impression of change. Risks are also assessed with adverse event collection.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Patients with chronic pain (more than 6 months)
* Patients with peripheral or central neuropathic pain, fibromyalgia, algoneurodystrophy

Exclusion Criteria:

* Patient under 18 years of age,
* Patient not requiring prescription of ketamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-07-07 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of benefit | At baseline
  Benefits (pain release after ketamine use) will be assessed by the Pain by the Numerical Pain Rating Scale (NPRS): the scale ranges from 0 no pain to 10 maximal tolerable pain, and risks will be assessed by collecting the ketamine adverse events reported by the patient and by the physician.

SECONDARY OUTCOMES:
Descriptive analysis of risk (by collecting adverse event) of ketamine use. | At baseline
  Biological statements will be collected during the usual care of patients, if possible (ASAT, ALAT, total bilirubin, conjugate bilirubin, free bilirubin, gamma glutamyl transferase, alkaline phosphatase,…)
Neuropathic Pain in 4 questions (DN4), | At baseline
  The Neuropathic pain in 4 questions (DN4) at baseline only. DN4 is a clinical tool for the diagnosis of neuropathic pain. This questionnaire has four questions divided into 10 items related to the interview (ie, symptoms) and to the sensory examination (ie, signs). The investigator asks and examines the patient and notes a response "no" or "yes" for each item: "yes" is scored as "1" and "no" is scored as "0". The sum of scores gives the total score of the patient (/10). DN4 is considered as positive if the patient obtains a score of 4/10.
Patient Global Impression of Change, the characteristics of pain (PGIC) | At baseline
  The Patient Global Impression of Change is a scale of global perception of change ("Deterioration" or "Improvement") realized at each telephone call except for baseline. This scale is graduated from 1 = very strongly improved to 7 = very strongly aggravated
Emotional status by Hospital Anxiety and Depression scale (HAD) | At baseline
  The HAD scale is a self-administered questionnaire in 14 items completed by the patient. It is used to determine the levels of anxiety and depression. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Global score ranges from 0 to 42.
Quality of life (Short Form 12 items Short Form survey) | At baseline
  assessed by a quality of life questionnaire (Short Form 12 items Short Form survey (SF12)

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Corriger A, Voute M, Lambert C, Pereira B, Pickering G; OKAPI Consortium. Ketamine for refractory chronic pain: a 1-year follow-up study. Pain. 2022 Apr 1;163(4):690-701. doi: 10.1097/j.pain.0000000000002403. PMID 34252909